CLINICAL TRIAL: NCT03303157
Title: REM Sleep and Dreaming- a Case Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Investigator, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-17-RT-0208-CTIL
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — not relevant

SUMMARY:
a case study of a man with a unique condition that negatively affects his sleep architecture. we want to study this man's sleep and see (through interviews) how his condition affects his ability to dream

ELIGIBILITY:
Inclusion Criteria:

- one patient- not relevant

Exclusion Criteria:

-

one patient- not relevant

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: one subject
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2017-11-20 (Estimated); Study Completion 2018-08-20 (Estimated)

PRIMARY OUTCOMES:
dream reports | 5 nights
  dream free-recall upon awakenings